CLINICAL TRIAL: NCT01478997
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group, Multi-Centric Study to Determine Whether Flexsure is Safe, Tolerable and Effective in Relieving Symptoms of Moderate Osteoarthritis of the Knee
Brief Title: A Study for Moderate Osteoarthritis of the Knee
Acronym: Flexsure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: VitalgNetics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA/110114/FLX/OA
Record Dates: First submitted 2011-11-17; First posted 2011-11-24 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexsure Capsules (Experimental): Investigational Product
  Interventions: Dietary Supplement: Flexsure Capsules
- Carboxy Methyl Cellulose Capsules (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: Flexsure Capsules — Flexsure - 3 capsules once a day in the absence of meals (at least 30 min prior to meals) for 56 days
  Other Names: Paracetamol
  Arms: Flexsure Capsules
Dietary Supplement: Placebo Capsules — Carboxy Methyl Cellulose
  Other Names: Paracetamol
  Arms: Carboxy Methyl Cellulose Capsules

SUMMARY:
This is a study to determine whether Flexsure is Safe, Tolerable and Effective in relieving symptoms of Moderate Osteoarthritis of the Knee.

DETAILED DESCRIPTION:
Primary efficacy variable:

Number of patients showing 20% reduction from baseline in the WOMAC - pain subscale

Secondary efficacy variables:

* Number of patients showing a 50% reduction from baseline in the WOMAC - pain subscale
* Number of patients showing a 20% reduction from baseline in VAS-pain
* Number of patients showing a 50% reduction from baseline in VAS- pain
* Mean change (percentage reduction) in WOMAC scores for pain, stiffness and physical function from baseline, as compared to placebo
* Mean change (percentage reduction) in VAS - pain, as assessed at clinic visits and by daily records in patient diary (First two weeks only)
* Consumption of rescue medication
* Investigator's Global assessment of efficacy
* Subject's global assessment of efficacy

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female patients aged 30-65 years, and diagnosed of OA of the knee according to the ACR clinical and radiographic criteria
* ARA functional class II or III
* Kellgren Lawrence radiological severity of Grade II, Grade III OA knee
* Maximal OA pain on movement, as measured on a 0-100 Visual analog scale (VAS) should be more than 40 and less than 80 in the previous 24 hrs at screening and baseline visits

Exclusion Criteria:

* Conditions that can mimic OA knee pain, E.g. rheumatoid arthritis, systemic lupus erythematosus, gout, psoriatic arthritis, pseudo gout or pain due to malignant disease
* BMI >35 kg/m2
* Indication of surgery for OA knee
* Arthroscopy of either knee in the past year
* Use of analgesics or any other symptom-relieving medication within 7 days of screening
* Use of systemic steroids or herbal medication for OA within 4 weeks of screening
* Use of Vit. D3 injections, Glucosamine sulphate, Chondroitin sulphate, Diacerin, Alendronate in the past 3 months
* Administration of intra-articular steroids in the past 3 month or hyaluronic acid in the last 9 months
* History of osteoporotic/ osteoarthritic fractures within the past 6 months
* Pregnant or lactating women or women with inadequate contraceptive measures
* Evidence or clinical suspicion of any major medical conditions (E.g. uncontrolled diabetes mellitus, uncontrolled hypertension, cardiovascular disease, thyroid, hepatic, renal dysfunction)
* Presence of any clinically significant laboratory anomaly
* Known cases of AIDS (HIV positive)
* History of Coronary Angioplasty/CABG within the past 2 years
* Moderate to severe peripheral neuropathy or other neurological disorders
* Alcohol abuse, medication or drug dependence
* Concurrent or previous participation in a clinical study within previous 6 weeks

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
WOMAC - pain subscale | 56 Days
Clinical Adverse Events | 56 Days
Laboratory Adverse Events | 56 Days
Assessment of Tolerability by the Subject | 56 Days

SECONDARY OUTCOMES:
Visual Analog Scale - Pain | 56 Days
Consumption of Rescue Medication | 56 Days
Investigator's and Subject's Global Assessment | 56 Days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Bhakti Shinde, BAMS, PGDCR, Study Chair — Vedic Lifesciences Pvt. Ltd.
Locations (2):
- India (2):
  - Nasik, Nashik, Maharashtra
  - Pune, Pune, Maharashtra